CLINICAL TRIAL: NCT07111273
Title: Diagnostic Value of Quantitative Fecal Immunochemical Test (qFIT) and Calprotectin (FC) Dynamic Changes at 2 Weeks for Predicting 52-Week Relapse or Treatment Escalation in Biologic-Naive Ulcerative Colitis: A Multicenter, Prospective Cohort Study (DYNAMIC-UC)
Brief Title: DYNAMIC-UC: Early qFIT and Calprotectin Change Predicting Relapse in Biologic-Naive Ulcerative Colitis
Acronym: DYNAMIC-UC
Status: Not yet recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Qilu Hospital of Shandong University (Qingdao) (Other); Dezhou Hospital Qilu Hospital of Shandong University (Other); JiNing NO.1 People Hospital (Unknown); Zaozhuang Municipal Hospital (Other); caoxian chinese medicine hospital (Unknown); longkou chinsese medicine hospital (Unknown); Shouguang people's Hospital (Unknown); Weihai Municipal Hospital (Other); Liaocheng People's Hospital (Other); ZhangQiu Yile Hospital (Unknown)
Responsible Party: Principal Investigator, Yan Zhang, MD, M.D, Qilu Hospital of Shandong University
Other Study IDs: QILUGI-001; QILUGILAB (Registry Identifier: DYNAMIC-UC)
Record Dates: First submitted 2025-07-30; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Ulcerative Colitis (UC); Fecal Calprotetin; FIT; Biomarker
Keywords: ulcerative colitis; fecal calprotectin; FIT; biologic-naive
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: FC and FIT TEST at WEEK0 2 4 — FC and FIT TEST at WEEK0 2 4

SUMMARY:
This multicenter prospective cohort study aims to evaluate whether a >50% decrease or normalization of both quantitative fecal immunochemical test (qFIT) and fecal calprotectin (FC) levels at 2 weeks after starting conventional therapy (mesalazine or corticosteroids) can predict clinical relapse or need for biologic/JAK inhibitor therapy escalation by 52 weeks in biologic-naive patients with active ulcerative colitis (UC). Secondary objectives include assessing predictive value at 4 weeks, building dynamic prediction models, conducting health economic evaluation (Number Needed to Test, NNT), and exploring baseline predictors of early biomarker response. Patients will be observed during standard care with stool samples collected at Weeks 0, 2, and 4. Biomarker results will be blinded to clinicians/patients until study completion.

DETAILED DESCRIPTION:
This is a prospective, observational cohort study conducted across multiple centers in China. Biologic-naive UC patients (Mayo Endoscopic Subscore ≥2) initiating conventional therapy (mesalazine or corticosteroids) will be enrolled. Stool samples for quantitative FIT (qFIT) and fecal calprotectin (FC) will be collected at Baseline (Week 0) , Week 2 (±3 days) , and Week 4 (±3 days) . Patients are classified at Week 2:

Group A (Rapid Responders): Both qFIT & FC decrease >50% from baseline OR normalize.

Group B (Slow/Non-Responders): Either qFIT or FC decrease ≤50%. The primary endpoint is the composite event rate (clinical relapse OR treatment escalation to biologics/JAK inhibitors) by Week 52 (±2 weeks) . Clinical relapse is defined as an increase ≥2 points in partial Mayo score (excluding endoscopy) with a rectal bleeding subscore ≥1 requiring therapy adjustment. Treatment escalation occurs per standardized criteria (steroid-refractoriness or dependence). Secondary endpoints include time-to-event, corticosteroid-free remission, mucosal healing at Week 52, predictive model performance (AUC, sensitivity, specificity), NNT calculation, and baseline predictors.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years.
* Established diagnosis of Ulcerative Colitis (UC) confirmed by clinical, endoscopic, and histopathological criteria.
* Endoscopic disease activity (Mayo Endoscopic Subscore ≥ 2) confirmed by colonoscopy during screening.
* Biologic-naive (no prior exposure to any biologic agent [e.g., infliximab, adalimumab, vedolizumab, ustekinumab] or JAK inhibitor).
* No use of systemic corticosteroids (oral or intravenous) within 4 weeks prior to Baseline (Week 0) visit.
* If using oral or rectal mesalazine/5-ASA preparations, dose must have been stable for ≥2 weeks prior to Baseline (Week 0).

Willing and able to provide written informed consent.

Exclusion Criteria:

* Diagnosis or high suspicion of Crohn's disease, ischemic colitis, infectious colitis, radiation colitis, intestinal tuberculosis, or other types of colitis.

Presence of other conditions clearly causing intestinal bleeding (e.g., acute hemorrhoidal bleeding, colorectal cancer, large colorectal polyps >1cm, intestinal vascular malformations).

* Untreated systemic conditions that may cause intestinal bleeding (e.g., thrombocytopenia [PLT <50 x 10^9/L], severe coagulopathy).
* Regular use of antiplatelet agents (e.g., aspirin, clopidogrel) or anticoagulants (e.g., warfarin, rivaroxaban).
* Pregnancy or lactation.
* Any other condition deemed by the investigator to make the patient unsuitable for study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ulcerative Colitis patints come to clinic or ward of hospitals.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Composite Endpoint Rate (Clinical Relapse OR Treatment Escalation) | From enrollment to Week 52 (±2 weeks)
  Proportion of patients experiencing either: 1) Clinical Relapse: Increase ≥2 points in partial Mayo Score (stool frequency + rectal bleeding + PGA) with rectal bleeding subscore ≥1 requiring therapy adjustment, OR 2) Treatment Escalation: Initiation of any biologic agent (e.g., infliximab, adalimumab, vedolizumab, ustekinumab) or JAK inhibitor due to steroid-refractoriness (failure to respond by Week 4) or steroid-dependence (relapse during/after steroid taper within 3 months) as per standardized protocol.

SECONDARY OUTCOMES:
Time to First Composite Endpoint Event | From enrollment to Week 52 (±2 weeks)
Proportion with Corticosteroid-Free Clinical Remission | Week 52 (±2 weeks)
  Partial Mayo Score ≤1 point without corticosteroid use for ≥4 weeks.
Diagnostic Performance (AUC) of Week 2 Biomarker Response | Week 2 prediction assessed at Week 52
  Area Under the Receiver Operating Characteristic Curve (AUC) for the Week 2 qFIT+FC combined response (Group A vs B) in predicting the Week 52 composite endpoint.
Number Needed to Test (NNT) | Week 52 (±2 weeks)
  NNT = 1 / [Event Rate (Group B) - Event Rate (Group A)] for the composite endpoint at Week 52.
Diagnostic Performance (AUC) of Biomarker Change Slope Models | Weeks 0-2 and Weeks 0-4 slopes assessed at Week 52
  AUC of logistic regression models using the rate of change (Δ/week) of FC and/or qFIT from Week 0 to Week 2 and/or Week 0 to Week 4 for predicting the Week 52 composite endpoint. Sensitivity, specificity, PPV, NPV will also be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided